CLINICAL TRIAL: NCT03240848
Title: Comparison of Artificial Intelligent Clinic and Normal Clinic for Diagnosing Congenital Cataracts
Brief Title: Comparison of Artificial Intelligent Clinic and Normal Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CCPMOH2017-China-5
Record Dates: First submitted 2017-07-30; First posted 2017-08-07 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Cataract
Keywords: congenital cataract; artificial intelligent clinic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Slit-lamp photography and patient recruitment will be performed in each participating clinic by trained clinical staffs. The clinical staffs, investigators involved in data management and analysis, and experts providing the gold standard diagnosis by consensus in each clinic will be blinded to the group assignment. The study participants, the coordinator, senior consultants, and study personnel responsible for randomisation will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial intelligent clinic (Experimental): Procedure: the initial diagnosis from artificial intelligent clinic Participants in group A assigned to artificial intelligent clinic to get the initial diagnosis after the eye examinations, including images of ocular anterior segment.
  Procedure: the final definite diagnosis from experts After making the initial diagnosis in artificial intelligent clinic, participants in group A went to get the final definite diagnosis from experts with more than 10 years of clinical experience.
  Interventions: Procedure: artificial intelligent clinic; Procedure: experts diagnose
- normal clinic (Active Comparator): Procedure: the initial diagnosis from normal clinic Participants in group B assigned to normal clinic to get the initial diagnosis after the eye examinations, including images of ocular anterior segment.
  Procedure: the final definite diagnosis from experts After making the initial diagnosis in normal clinic, participants in group B went to get the final definite diagnosis from experts with more than 10 years of clinical experience.
  Interventions: Procedure: normal clinic; Procedure: experts diagnose

INTERVENTIONS:
Procedure: artificial intelligent clinic — Participants in group A assigned to artificial intelligent clinic to get the initial diagnosis after the eye examinations, including images of ocular anterior segment.
  Arms: artificial intelligent clinic
Procedure: normal clinic — Participants in group B assigned to normal clinic to get the initial diagnosis after the eye examinations, including images of ocular anterior segment.
  Arms: normal clinic
Procedure: experts diagnose — After making the initial diagnosis, participants went to get the final definite diagnosis from experts with more than 10 years of clinical experience.

SUMMARY:
In this study, the investigators provide participants≤14 years old the artificial intelligent clinic or normal clinic in the purpose of seeking out a better way to make a definite diagnosis with high efficiency and accuracy, and report a prospective, randomized controlled study aiming at comparison of artificial intelligent clinic and normal clinic for diagnosing congenital cataract.

DETAILED DESCRIPTION:
Children ≤14 years old from ophthalmic clinic without treatment were enrolled to a prospective, randomized controlled study. Patients were assigned to two groups: participants in group A went to the artificial intelligent clinic and get the initial diagnosis, while in Group B, the participants went to the normal clinic. Investigators provide the final definite diagnosis from experts for two groups. Investigators compared the accuracy of the diagnosis, time consuming and the satisfaction level between two groups, aiming at comparison of artificial intelligent clinic and normal clinic for diagnosing congenital cataract.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients from collaborating eye clinics Written informed consents provided

Exclusion Criteria:

* Definitive diagnosis of cataract or other ocular abnormalities Previous eye surgery Can not cooperate with the slip lamp examination Unwilling to participate in this trail

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
The accuracy of artificial intelligence diagnosis for congenital cataract | baseline
  The accuracy of artificial intelligence diagnosis was calculated.

SECONDARY OUTCOMES:
The evaluation of disease severity and treatment determination | baseline
  The accuracy of the evaluation of disease severity and treatment determination was calculated
The time consuming of diagnosis | baseline
  The time consuming of diagnosis was calculated.
The level of patients' satisfaction | baseline
  The information about patients' satisfaction was recorded by using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin H, Li R, Liu Z, Chen J, Yang Y, Chen H, Lin Z, Lai W, Long E, Wu X, Lin D, Zhu Y, Chen C, Wu D, Yu T, Cao Q, Li X, Li J, Li W, Wang J, Yang M, Hu H, Zhang L, Yu Y, Chen X, Hu J, Zhu K, Jiang S, Huang Y, Tan G, Huang J, Lin X, Zhang X, Luo L, Liu Y, Liu X, Cheng B, Zheng D, Wu M, Chen W, Liu Y. Diagnostic Efficacy and Therapeutic Decision-making Capacity of an Artificial Intelligence Platform for Childhood Cataracts in Eye Clinics: A Multicentre Randomized Controlled Trial. EClinicalMedicine. 2019 Mar 17;9:52-59. doi: 10.1016/j.eclinm.2019.03.001. eCollection 2019 Mar. PMID 31143882